CLINICAL TRIAL: NCT01624064
Title: A Double Blind Clinical Trial to Examine the Renal Effects of an Angiotensin Converting Enzyme Inhibitor (Enalapril) in Adults With Chronic Kidney Disease of Uncertain Aetiology (CKDu)
Brief Title: Renal Effects of an Angiotensin Converting Enzyme Inhibitor in Adults With Chronic Kidney Disease of Uncertain Aetiology
Acronym: CKDu
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ministry of Health, Sri Lanka (Other Government)
Collaborators: World Health Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NSF CKDu Research
Record Dates: First submitted 2012-06-16; First posted 2012-06-20 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-06

CONDITIONS: Renal Insufficiency, Chronic
Keywords: Renal Insufficiency, Chronic; Uncertain aetiology; ACEI
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Enalapril; Angiotensin-Converting Enzyme Inhibitors; calcium lactate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Enalapril, Proteinuria < 1g/day (Active Comparator)
  Interventions: Drug: Enalapril
- Calcium, Proteinuria < 1g/day (Placebo Comparator)
  Interventions: Drug: Calcium Supplement
- Enalapril, Proteinuria > 1g/day (Active Comparator)
  Interventions: Drug: Enalapril
- Calcium, Proteinuria > 1g/day (Placebo Comparator)
  Interventions: Drug: Calcium Supplement

INTERVENTIONS:
Drug: Enalapril — 2.5-20 mg/day
  Other Names: Angiotensin Converting Enzyme Inhibitor
  Arms: Enalapril, Proteinuria < 1g/day; Enalapril, Proteinuria > 1g/day
Drug: Calcium Supplement — Calcium 2.5-20 mg/day
  Other Names: Calcium lactate
  Arms: Calcium, Proteinuria < 1g/day; Calcium, Proteinuria > 1g/day

SUMMARY:
Enalapril would significantly reduce progression of renal disease in patients with Chronic Kidney Disease of Uncertain aetiology.

DETAILED DESCRIPTION:
End Stage Kidney Disease (ESKD) results in reduced life expectancy, quality of life and increased consumption of health care resources. Chronic Kidney Disease of Uncertain aetiology (CKDu) is being increasingly recognized in the North Central Region of Sri Lanka and in certain regions over 25% (unpublished data) of general population is suspected as suffering from CKDu. The number of patients who reach ESKD that requires hemodialysis or transplantation is increasing, highlighting the need to find strategies that slow progression of kidney disease. The need for these strategies is even more critical in Sri Lanka where dialysis in not a preferred treatment option. Treatment strategies should be readily accessible and cheap.

The importance of proteinuria as a significant risk factor for ESKD is well recognized, and treatment that is targeted at reducing proteinuria has been shown to reduce progression of renal disease. The Renin - Angiotensin - Aldosterone - System (RAAS) is directly involved in the regulation of blood pressure, fluid volume, and vascular response to injury and inflammation. The inappropriate activation of this system causes hypertension, fluid retention, and inflammatory, thrombotic, and atherogenic effects that may contribute to end-organ damage in the long term. Angiotensin II mediates hemodynamic effects as well as inflammation and fibrosis in the kidney, heart, and vasculature.

Numerous clinical trials have established that interruption of the RAAS cascade with angiotensin-converting enzyme inhibitors (ACEI) or angiotensin receptor blockers (ARB) is beneficial in slowing progression of renal disease. Reduction of BP lowers proteinuria, but the use of an ACEI or an ARB reduces both proteinuria and the rate of deterioration of renal function beyond those seen with equivalent BP reduction from conventional antihypertensive agents. However, the use of these agents has limitations, with significant numbers of treated patients still demonstrating progressive renal disease. RAAS blockers have been shown to blunt the progression of advanced kidney disease. However the long-term renal effect of these agents in early renal disease is not well demonstrated. In fact the trials which showed benefits with RAAS blockers did show in glomerular disease and evidence is not so strong in tubulo-interstitial disease. The benefits of RAS inhibition seem to depend on the degree of proteinuria at baseline. It is marginal in those with low grade proteinuria.

In most forms of proteinuric chronic renal disease, glomerular filtration rate continues to decline even when the initial insult has been removed. The cause of CKDu is still unknown. CKDu is a tubulo-interstitial disease with low grade proteinuria. We believe that the place of ACEI for secondary prevention of CKDu progression needs investigation

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 18-70 years of age
* CKDu Grade 1, 2, 3
* No contraindication for treatment with ACEI
* Informed consent given

Exclusion Criteria:

* Grade 4 CKDu
* Other chronic diseases
* Evidence or suspicion of non renal secondary hypertension
* Diabetes type 1 or 2
* Evidence or suspicion of renovascular disease, obstructive uropathy, or other renal disease
* Treatment with corticosteroids, non-steroidal anti-inflammatory drugs, or immune-suppressive drugs
* Acute myocardial infarction or cerebrovascular accident in the previous 6 months
* Severe uncontrolled hypertension (diastolic blood pressure ≥115 and/or systolic blood pressure ≥220 mm Hg)
* Suspicion or evidence of connective tissue disease, cancer, higher serum aminotransferase concentrations
* Chronic cough; drug or alcohol abuse; pregnancy and breast feeding
* Unwillingness to sign informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-08; Primary Completion 2012-10 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Proteinuria | One year
  Numerous clinical trials have established that angiotensin-converting enzyme inhibitors (ACEI) are beneficial in slowing progression of renal disease. However the long-term renal effect of these agents in early renal disease is not well demonstrated. In fact the trials which showed benefits with ACEI did show in glomerular disease and evidence is not so strong in tubulo-interstitial disease.
Estimated GFR | One year
  In most forms of proteinuric chronic renal disease, glomerular filtration rate continues to decline even when the initial insult has been removed. The cause of CKDu is still unknown. CKDu is a tubulo-interstitial disease with low grade proteinuria. We believe that the place of ACEI for secondary prevention of CKDu progression needs investigation.

SECONDARY OUTCOMES:
All cause mortality | One year
Cardiovascular mortality | One year

CONTACTS AND LOCATIONS:
Overall Officials: Selvarajah Mathu, MBBS, MD, Principal Investigator — Ministry of Health; Shanthi Mendis, MBBS, MD, Principal Investigator — World Health Organization; Rezvi Sheriff, MBBS, MD, Principal Investigator — University of Colombo; Thilak Abeysekera, MBBS, MD, Principal Investigator — Ministry of Health; Saroj Jayasinghe, MBBS, MD, Principal Investigator — University of Colombo
Locations (1):
- General (Teaching) Hospital, Anuradhapura, Anuradhapura, North Central Province, Sri Lanka